CLINICAL TRIAL: NCT01755741
Title: A Multicenter, Open-Label, Randomized, Two-Period, Crossover Non-inferiority Trial to Assess the Functionality of Male Condoms With a Silicone Elastomer Vaginal Ring
Brief Title: Functionality of Male Condoms With a Silicone Elastomer Vaginal RIng
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: International Partnership for Microbicides, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: IPM 029
Record Dates: First submitted 2012-11-27; First posted 2012-12-24 (Estimated); Last update posted 2018-03-29 (Actual); Status verified 2018-03

CONDITIONS: Human Immunodeficiency Virus
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Condoms

STUDY DESIGN:
Intervention Model Description: IPM 029 is an open-label, randomized, two-period, crossover non-inferiority trial conducted at two research centers in the U.S. to assess condom functionality during vaginal intercourse in healthy, monogamous heterosexual, sexually active couples.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo Vaginal Ring (Experimental): Placebo vaginal ring with condom use
  Interventions: Combination Product: Placebo Vaginal Ring; Device: Condom
- Condom (Other): Male condoms during vaginal intercourse in presence and absence of the vaginal ring.
  Interventions: Device: Condom

INTERVENTIONS:
Combination Product: Placebo Vaginal Ring — a silicone elastomer placebo vaginal ring, similar in composition to the dapivirine Ring-004 (which is currently used in IPM's ongoing Phase III program), except that it did not contain any active pharmaceutical agent, and a commercially available standard male latex condom with a silicone-based lubricant.
  Arms: Placebo Vaginal Ring
Device: Condom — Male condom

SUMMARY:
This trial will assess the potential impact of a vaginal ring on condom use by comparing the performance (total clinical failure, clinical slippage, and clinical breakage) of a standard male lubricated latex condom when the female partner is wearing the vaginal ring and when the female partner is not wearing the vaginal ring.

ELIGIBILITY:
Inclusion Criteria:

1. Mutually monogamous heterosexual couples; current relationship ≥3 months; and who can give written informed consent;
2. Age ≥18 to ≤45 years (females) or ≥18 to ≤55 years (males) at time of the screening visit;
3. Healthy on the basis of medical history;
4. Not at risk of pregnancy, i.e., female is surgically sterile, using an IUD, or using effective hormonal contraception, or has a vasectomized partner. The use of vaginal contraceptive rings will not be allowed;
5. Sexually active and agree to have at least 8 acts of penile-vaginal intercourse using a study condom over 2 periods of up to 4 weeks each;
6. Agree to use only the condoms provided by trial personnel during the time of participation. Additional lubricant will be provided; use of non-study lubricants will not be allowed;
7. Agree to not use other vaginal products, except menstrual absorption products (e.g. tampons) and study lubricant during the trial;
8. Available for all visits and consent to follow all procedures scheduled for the trial;
9. At low risk for HIV infection.

Exclusion Criteria:

1. Males with untreated erectile dysfunction;
2. Female with positive pregnancy test;
3. Either partner allergic to natural latex or vaginal lubricants such as Astroglide ®;
4. History by self-report of recurrent or a recently-treated (within past 2 weeks) sexually transmitted infection (e.g. gonorrhea, syphilis, chlamydia) or HIV(+);
5. Currently using condoms for protection against sexually transmitted infection;
6. Either partner taking any topical or oral medication to treat a urogenital condition at enrollment, except medication for the male partner to treat erectile dysfunction (e.g., tadalafil, sildenafil);
7. Either partner with a self-reported or clinically diagnosed urogenital condition (e.g. itching, burning, irritation, etc.) that, in the opinion of the Investigator, could affect use of the study condoms or ability to interpret trial data;
8. Females, based on findings from a pelvic examination, who are not suitable candidates for wearing the vaginal ring (anatomical condition, current vaginal infection, etc.);
9. Current participation in a study or other research involving a drug, device or other product;
10. Any condition(s) that, in the opinion of the Investigator, might interfere with adherence to trial requirements or evaluation of the trial objectives.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2013-02; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Total clinical failure rate (N slipped or broken/N total) off the penis or broke during intercourse or withdrawal, divided by the number of condoms used during intercourse. | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ron Frezieres, Principal Investigator — California Family Health Council
Locations (2):
- United States (2):
  - California Family Health Council, Berkeley, California
  - California Family Health Council, Los Angeles, California

IPD SHARING:
Plan to Share IPD: No